CLINICAL TRIAL: NCT00760201
Title: Analysis of Hospital Executives, Physician Administrators, and Hospital Legal Counsels� Perceptions of End-of-Life Care
Brief Title: Qualitative Analysis of Hospital Executives, Physician Administrators, and Hospital Legal Counsels' Perceptions of End-of-Life Care
Acronym: HospExe
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Garner, Kimberly - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 9360
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: End of Life Care
Keywords: executive; administrator; perceptions; legal counsel; end of life
MeSH Terms: conditions — Death

STUDY DESIGN:
Biospecimen Retention: Qualitative Analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Hospital executives, physician administrators and hospital legal counsel

SUMMARY:
Interviewing hospital executives, physician administrators and hospital legal counsel who work in a hospital setting (academic, governmental, private or community hospital) about their perceptions concerning current and future end-of-life care provided in their facilities

ELIGIBILITY:
Inclusion Criteria:

Informant is a hospital executive, physician administrator or hospital legal counsel in a hospital setting (academic, governmental, private or community hospital) and is able to communicate perceptions verbally through use of English language. All participants will likely be nonveterans

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hospital executive, physician administrator or hospital legal counsel in a hospital setting (academic, governmental, private or community hospital)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Perceptions of hospital executive, physician administrator or hospital legal counsel in a hospital setting (academic, governmental, private or community hospital) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly K. Garner, MD JD MPH, Principal Investigator — Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock
Locations (1):
- Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas, United States